CLINICAL TRIAL: NCT05497804
Title: REsponse Adapted Combination Therapy Approaches for High-Risk Multiple Myeloma (REACH)
Brief Title: Combination Treatment Therapy Approaches for the Treatment of High-Risk Multiple Myeloma, REACH Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC210811; P50CA186781 (NIH); NCI-2022-06150 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-002687 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-08-03; First posted 2022-08-11 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: ISS Stage III Plasma Cell Myeloma; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Biopsy; carfilzomib; daratumumab; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Lenalidomide; Magnetic Resonance Spectroscopy; Specimen Handling; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (combination chemotherapy) (Experimental): INDUCTION: Patients receive carfilzomib IV on days 2, 8, and 15 of cycle 1 and days 1, 8, and 15 of cycles 2-12, lenalidomide PO days 1-21 of each cycle, daratumumab SC days 1, 8, 15, and 22 of cycles 1 and 2, days 1 and 15 of cycles 3-6, and day 1 of subsequent cycles, and dexamethasone PO or IV on days 1, 8, 15, and 22 of each cycle. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients receive carfilzomib IV on days 1, 8, and 15, lenalidomide PO days 1-21, daratumumab SC day 1 of each cycle. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive carfilzomib IV on day 1, lenalidomide PO days 1-21, daratumumab day 1 of each cycle. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspirate and biopsy, MRI and, CT/PET.
  Interventions: Procedure: Bone Marrow Aspiration and Biopsy; Drug: Carfilzomib; Procedure: Computed Tomography; Biological: Daratumumab; Drug: Dexamethasone; Drug: Lenalidomide; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Multigated Acquisition Scan; Procedure: Biospecimen Collection; Procedure: Echocardiography; Procedure: Chest Radiography

INTERVENTIONS:
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration and biopsy
Drug: Carfilzomib — Given IV
  Other Names: Kyprolis; PR-171
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Biological: Daratumumab — Given SC
  Other Names: Darzalex; HuMax-CD38; JNJ-54767414; Daratumumab Biosimilar HLX15; Daratumumab-fihj
Drug: Dexamethasone — Given IV/PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Procedure: Chest Radiography — Undergo chest x-ray
  Other Names: chest x-ray

SUMMARY:
This phase II trial test whether combination chemotherapy works to improve blood test results in patients with high-risk multiple myeloma. Chemotherapy drugs, such as carfilzomib, daratumumab, lenalidomide, and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. This trial may help determine if patients who have a small amount of cancer left after the initial treatment, called minimal residual disease, will benefit from the drug combination.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the rate of sustained minimal residual disease (MRD) negativity (MRD negative status at any point, with a repeated MRD negative status one year later) in subjects with high-risk multiple myeloma.

SECONDARY OBJECTIVES:

I. To describe the toxicities associated with this treatment approach in subjects with high-risk multiple myeloma (MM).

II. To estimate the overall response rate, very good partial response (VGPR) or better rate and complete response (CR) rate at the end of induction, end of consolidation, end of maintenance and at two years after the completion of treatment.

III. To estimate the progression-free survival and overall survival rate.

CORRELATIVE RESEARCH OBJECTIVES:

I. To describe the clonal architecture through a combination of genomic, epigenomic, proteomic and metabolomic studies before and after treatment, in subjects with high-risk MM.

II. To describe the bone marrow microenvironment through various stages of treatment and the time of MRD negative state and at time of relapse.

OUTLINE:

INDUCTION: Patients receive carfilzomib intravenously (IV) on days 1, 2, 8, and 15 of cycle 1 and days 1, 8, and 15 of cycles 2-12, lenalidomide orally (PO) days 1-21 of each cycle, daratumumab subcutaneously (SC) days 1, 8, 15, and 22 of cycles 1 and 2, days 1 and 15 of cycles 3-6, and day 1 of subsequent cycles, and dexamethasone PO or IV on days 1, 8, 15, and 22 of each cycle. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Patients receive carfilzomib IV on days 1, 8, and 15, lenalidomide PO days 1-21, daratumumab SC day 1 of each cycle. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive carfilzomib IV on day 1, lenalidomide PO days 1-21, daratumumab SC day 1 of each cycle. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity.

Additionally, patients undergo bone marrow aspirate and biopsy, blood sample collection, echocardiography (ECHO) or multigated acquisition (MUGA) scan, and magnetic resonance imaging (MRI), computed tomography (CT), or positron emission tomography (PET)/CT throughout the study. Patients also undergo chest radiography (x-ray) during screening.

After completion of study treatment, patients are followed up every 6 months for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION-INCLUSION CRITERIA:
* Age >= 18 years and =< 80 years.
* Patient must have suspected or confirmed newly diagnosed multiple myeloma by International Myeloma Working Group (IMWG) criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
* Provide informed written consent.
* Willing to return to enrolling institution for follow-up during the active treatment phase of the trial.
* Willing to provide blood and bone marrow samples for planned research.
* Life expectancy > 6 months.
* Able to take aspirin (325 mg) daily as prophylactic anticoagulation.

  * Note: subjects intolerant to aspirin may use warfarin, novel oral anticoagulants, or low dose molecular weight heparin.
* Patients must have monoclonal protein studies (serum free light chain assay, serum immunofixation or serum matrix-assisted laser desorption ionization time-of-flight mass-spectrometry [MASS-FIX]) at time of diagnosis before induction therapy initiated and available for review to be enrolled. Note: Patients are allowed to participate in this study if urine electrophoresis immunofixation study was not done at time of diagnosis or cannot be obtained
* REGISTRATION-INCLUSION CRITERIA:
* High risk myeloma, which is untreated, defined as any two of:

  * Beta-2 microglobulin >5.5
  * Gain or amplification of chr1q
  * del17p or monosomy 17 or TP53 mutation (if known)
  * t(4;14) or t(14;16)
  * >= 5% circulating plasma cells
  * presence of extramedullary disease (does not include bone contiguous disease)
* Creatinine clearance >= 30 mL/min (using Cockroft-Gault equation) (obtained =< 14 days prior to registration).
* Absolute neutrophil count (ANC) >= 1000/mm^3 (without the use of growth factors) (obtained =< 14 days prior to registration).
* Platelet count >= 75000/mm^3 (obtained =< 14 days prior to registration).
* Hemoglobin >= 8.0 g/dL.
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 14 days prior to registration).
* Alanine transaminase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN (obtained =< 14 days prior to registration).
* Registration must be completed =< 30 days after pre-registration.
* Patients must not have received more than one cycle of treatment between pre-registration and registration.
* All 4 drugs in the study regimen approved by insurance.
* Left ventricular ejection fraction (LVEF) >= 40% =< 30 days prior to pre-registration

Exclusion Criteria:

* PRE-REGISTRATION EXCLUSION:
* Monoclonal gammopathy of undetermined significance (MGUS), smoldering myeloma, light chain amyloidosis with organ involvement.
* Diagnosed or treated for another malignancy =< 1 year prior to pre- registration or previously diagnosed with another malignancy and have any evidence of residual disease.

  * NOTE: Subjects with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Other co-morbidity which would interfere with subject's ability to participate in trial, e.g. uncontrolled infection, uncompensated heart or lung disease.
* Other concurrent chemotherapy, or any ancillary therapy considered investigational. NOTE: Concurrent chemotherapy is any treatment not related to multiple myeloma.

  * NOTE: Concurrent chemotherapy is any treatment not related to multiple myeloma
  * NOTE: Bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment.
* Peripheral neuropathy >= grade 3 on clinical examination or grade 2 with pain =< 30 days prior to registration.
* Major surgery =< 14 days prior to pre-registration.
* Any medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Known allergies, hypersensitivity, or intolerance to corticosteroids, monoclonal antibodies or human proteins, or their excipients (refer to respective package inserts or investigator's brochure) or known sensitivity to mammalian-derived products. Known allergies, hypersensitivity, or intolerance to trial drugs.
* Inability to comply with protocol/procedures.
* Received prior treatment for multiple myeloma prior to pre-registration. Note: results can still be pending as long as the tests have been performed
* REGISTRATION-EXCLUSION CRITERIA:
* If any of the following exist at screening, subject will not be eligible for trial because this trial involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception (per protocol).
* Evidence of current uncontrolled cardiovascular conditions, including hypertension, cardiac arrhythmias, congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.

  * Note: Prior to trial entry, any electrocardiogram (ECG) abnormality at screening must be documented by the investigator as not medically relevant.
* New York Heart Association (NYHA) II, III, IV heart failure.
* Known human immunodeficiency virus (HIV) positive.
* Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie., subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels. Those who are PCR positive will be excluded.

  * EXCEPTION: subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
* Known or suspected active hepatitis C infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2027-11-20 (Estimated); Study Completion 2028-11-20 (Estimated)

PRIMARY OUTCOMES:
Rate of sustained minimal residual disease (MRD) negativity | At 1 year
  MRD negative status at any point, with a repeated MRD negative status one year later. All subjects meeting the eligibility criteria who have signed a consent form and have begun treatment will be evaluable, with the exception of subjects determined to be a major violation.

SECONDARY OUTCOMES:
Overall response rate (>= confirmed very good partial response ([VGPR]) | End of induction, end of consolidation, and every 3 cycles of maintenance, up to two years or 24. One cycle is 28 days. after treatmentmonths
  Exact binomial 95% confidence intervals for the true response proportion at each time point will be calculated.
Overall survival | Up to 10 years
  Defined as the time from registration to death due to any cause. The distribution of overall survival will be estimated using the method of Kaplan-Meier.
Progression-free survival | Up to 10 years
  Defined as the time from registration to the earliest date of documentation of disease progression or death due to any cause. The distribution of progression-free survival will be estimated using the method of Kaplan-Meier.
Incidence of adverse events | Up to 30 days after administration of study therapy
  Adverse Events: All eligible subjects that have initiated treatment will be considered evaluable for assessing adverse event rate(s). The maximum grade for each type of adverse event will be recorded for each subject, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the trial treatment will be taken into consideration. AEs will be summarized overall, as well as by treatment phase (induction, consolidation, maintenance with carfilzomib and lenalidomide and daratumumab).

OTHER OUTCOMES:
Clonal architecture before treatment | Before and after treatment, up to two years or 24 months
  To determine the clonal architecture before treatment, after treatment in subjects with residual disease and in subjects who have disease progression after attaining MRD negativity.
Bone marrow microenvironment | Before and after treatment, up to two years or 24 months
  To evaluate the bone marrow microenvironment before and after treatment and the time of MRD negative state.

CONTACTS AND LOCATIONS:
Overall Officials: Shaji K. Kumar, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials